CLINICAL TRIAL: NCT03012178
Title: Prospective Evaluation of MRI as a Predictor of Outcomes in Patients Undergoing Mitral Valve Surgery: MRI-MVS Study
Brief Title: MRI as a Predictor of Outcomes in Patients Undergoing Mitral Valve Surgery
Acronym: MRI-MVS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 967510-2
Record Dates: First submitted 2016-12-16; First posted 2017-01-06 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Mitral Valve Insufficiency
Keywords: Mitral Regurgitation; Mitral valve Surgery; MRI
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mitral Valve Surgery: Patients undergoing ACC/AHA guideline directed mitral valve surgery for mitral insufficiency.
  Interventions: Procedure: Mitral valve surgery

INTERVENTIONS:
Procedure: Mitral valve surgery — ACC/AHA guideline directed mitral valve repair or replacement

SUMMARY:
Based on the ACC/AHA guidelines for the management of mitral valve disease, quantifying the severity of mitral regurgitation is central to determining which patients are appropriate for correction of their mitral valve by surgery. Specifically, once the diagnosis of severe MR is made, patients are considered appropriate for mitral valve surgery in almost all clinical circumstances. However, there is a significant mortality and morbidity associated with mitral valve surgery The most common diagnostic tool to assess the severity of MR is echocardiography. Several studies have shown that echocardiography parameters used to quantify and qualify MR have high inter-observer and intra-observer variability, calling the accuracy of these parameters into question. Furthermore, studies have shown that there is a significant degree of discordance between echocardiography and MRI when assessing MR, particularly among patients referred for mitral valve surgery. In a recent study, quantification of mitral regurgitant volume MRI was found to be more accurate than echocardiography in patients who underwent mitral valve surgery. All 38 patients who underwent mitral valve surgery in this study were deemed appropriate according the ACC/AHA guidelines based on echocardiographic findings. However, more than 2/3rds of patients who underwent mitral valve surgery in this study did not have severe MR by MRI. Thus, we propose this prospective multicenter trial to assess: 1) the severity of MR by MRI in patients undergoing mitral valve surgery. 2) the impact of mitral valve surgery on quality of life and healthcare costs in the context of MR severity by MRI, 3) assess patient outcomes post surgery in the context of MR severity by MRI and 4) the likelihood of valve replacement vs. repair according to MR severity by MRI.

DETAILED DESCRIPTION:
Mitral regurgitation is a common disease which can lead to heart failure and death if left untreated. The only known therapy for mitral regurgitation is correction of the mitral valve, most commonly performed by surgical repair or replacement. According the STS database, there were 15,748 lone mitral valve surgeries in 2014. The number of mitral valve surgeries has been increasing with a 23% increase between the years 2010 and 2014. Based on the ACC/AHA guidelines for the management of mitral valve disease, quantifying the severity of mitral regurgitation is central to determining which patients are appropriate for correction of their mitral valve by surgery. Specifically, once the diagnosis of severe MR is made, patients are considered appropriate for mitral valve surgery in almost all clinical circumstances. However, there is a significant mortality and morbidity associated with mitral valve surgery. In the STS database, 30 day mortality was ~2% for repair and ~5% for replacement. This data does not take into account long-term mortality and morbidity from re-operation and life-long anti-coagulation as well as changes in quality of life.

The most common diagnostic tool to assess the severity of MR is echocardiography. Several studies have shown that echocardiography parameters used to quantify and qualify MR have high inter-observer and intra-observer variability, calling the accuracy of these parameters into question. Furthermore, studies have shown that there is a significant degree of discordance between echocardiography and MRI when assessing MR, particularly among patients referred for mitral valve surgery. In a recent study, quantification of mitral regurgitant volume MRI was found to be more accurate than echocardiography in patients who underwent mitral valve surgery. All 38 patients who underwent mitral valve surgery in this study were deemed appropriate according the ACC/AHA guidelines based on echocardiographic findings. However, more than 2/3rds of patients who underwent mitral valve surgery in this study did not have severe MR by MRI. Thus, we propose this prospective multicenter trial to assess: 1) the severity of MR by MRI in patients undergoing mitral valve surgery. 2) the impact of mitral valve surgery on quality of life and healthcare costs in the context of MR severity by MRI, 3) assess patient outcomes post surgery in the context of MR severity by MRI and 4) the likelihood of valve replacement vs. repair according to MR severity by MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* Able to give informed consent.
* Undergoing lone mitral valve surgery for chronic primary mitral regurgitation within 30 days.
* Indication for mitral valve surgery is a class I or IIa according to the 2014 ACC/AHA guidelines for the management of valvular heart disease.

Exclusion Criteria:

* Secondary mitral regurgitation.
* Have a device which is not compatible with MRI
* Claustrophobia preventing MRI.
* Concomitant CABG, other valve surgery, or other cardiac surgery.
* Atrial fibrillation or other substantial arrhythmia that would substantially degrade MRI image acquisition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are scheduled to undergo ACC/AHA guideline directed mitral valve surgery for mitral regurgitation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Operative and peri-operative outcomes according to the mitral regurgitation severity quantified by MRI. | 2 years
  Operative and peri-operative outcomes (mortality, morbidity, hospitalizations, reoperation, bleeding, and CVA) in the context of mitral regurgitation severity quantified by MRI.

SECONDARY OUTCOMES:
Quality of life | 2 years
  Operative and peri-operative outcomes (mortality, morbidity, hospitalizations, reoperation, bleeding, and CVA) in the context of mitral regurgitation severity quantified by MRI.
Repair vs Replacement | 4 months
  Assess if the likelihood of mitral valve repair vs. replacement is associated with mitral regurgitant severity as quantified by MRI.
Severity of mitral regurgitation as quantified MRI in subjects who are undergoing guideline directed mitral valve surgery. | 0 days
  Cross sectional data regarding severity of mitral regurgitation as quantified MRI in subjects who are undergoing guideline directed mitral valve surgery
Correlation of pre-surgical regurgitant volume as quantified by MRI with post-surgical change in LV EDV. | 4 months
  Correlation of pre-surgical regurgitant volume as quantified by MRI with post-surgical change in LV EDV.

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown Medical Center, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uretsky S, Gillam LD, Biederman RWW, Han Y, Jacob R, Martin ET, Langer M, Choi AD, Sultan I, Cavalcante JL, Shah DJ, Tong MS, Wolff SD, Sakul S, Guglielmo M, Pontone G. Sex differences in pre- and post-surgical left ventricular remodelling and outcomes in primary mitral regurgitation. Eur Heart J Cardiovasc Imaging. 2025 Jul 31;26(8):1429-1437. doi: 10.1093/ehjci/jeaf151. PMID 40392571